CLINICAL TRIAL: NCT04830358
Title: A Single Center, Randomized, Single-blind, Active Comparator Phase 1 Clinical Trial to Assess the Safety and Immunogenicity of the 'EuPCV15' in Healthy Korean Adults
Brief Title: Safety and Immunogenicity of the 'EuPCV15' in Healthy Korean Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EuBiologics Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EuVCT_PCV101
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-03

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EuPCV15 (Experimental): Single dose of Pneumococcal Conjugate Vaccine will be administered intramuscularly at Day 0.
  Interventions: Biological: EuPCV15
- Prevenar13 (Active Comparator): Single dose of Pneumococcal Conjugate Vaccine will be administered intramuscularly at Day 0.
  Interventions: Biological: Prevenar13

INTERVENTIONS:
Biological: EuPCV15 — 15-valent Pneumococcal conjugate vaccine
  Arms: EuPCV15
Biological: Prevenar13 — 13-valent Pneumococcal conjugate vaccine
  Arms: Prevenar13

SUMMARY:
The safety and immunogenicity of EuPCV15 compared to Prevenar13 are assessed in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 19 to 50 years old
2. Participants willing to give written informed consent to participate in the trial

Exclusion Criteria:

1. History of invasive pneumococcal infection within 5 years at screening
2. Known hypersensitivity to any component of the study vaccine
3. Immune deficiency or immunosuppressive disorder
4. Immunized with any licensed vaccine within 4 weeks prior to screening
5. Pregnant, lactating women or women of childbearing age not using a reliable method of contraception
6. Participants who in the opinion of the investigator will not be able to comply with any of the protocol required procedure

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Solicited AEs (Local and Systemic) | within 14 days after vaccination
Incidence of Unsolicited AEs | within 28 days after vaccination
Incidence of SAEs | within 180 days after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Seoul St.Mary's Hospital, Seoul, South Korea